CLINICAL TRIAL: NCT06973213
Title: The Effect of Core Stabilization Exercises on Upper Extremity Function and Balance in Children With Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Core Stabilization for Upper Extremity Function and Balance in Children With Cerebral Palsy
Acronym: CORE-CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Çiğdem Çekmece, Assist. Prof. Dr., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KAEK/01.b1.02; E-66175679-514.13.02-1407423 (Other: Turkish Medicines and Medical Devices Agency)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy (CP); Upper Extremity Function; Core Stabilization Exercise Therapy; Balance; Trunk Stability
Keywords: cerebral palsy; upper extremity function; core stabilization exercises; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- intervention (Active Comparator)
  Interventions: Other: core exercises

INTERVENTIONS:
Other: core exercises — the intervention group underwent approximately 45 minutes of core stabilization exercises daily.
  Arms: intervention

SUMMARY:
This study investigates the effects of core stabilization exercises on balance and upper extremity function in children with cerebral palsy (CP). A total of 36 children aged 5 to 12 years with CP were randomly assigned to either an intervention group or a control group. Both groups received standard physiotherapy, rehabilitation, and occupational therapy five days a week for four weeks. In addition, the intervention group performed daily core stabilization exercises for approximately 45 minutes. The study assessed balance using the Pediatric Berg Balance Scale and the Trunk Control Measurement Scale, and upper extremity function using the Box and Block Test and the Assisting Hand Assessment before and after the treatment period.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of permanent disorders of movement and posture that occur due to non-progressive disturbances in the developing fetal or infant brain. Children with CP often experience deficits in trunk control, balance, and upper extremity function, which significantly affect their daily activities and quality of life. Core stabilization exercises are widely used in neurorehabilitation to improve trunk control and postural stability, potentially enhancing balance and upper limb function.

This randomized controlled trial aimed to evaluate the effects of core stabilization exercises on upper extremity function and balance in children with CP. The study included children aged 5 to 12 years, classified at levels I-III according to the Gross Motor Function Classification System (GMFCS) and the Manual Ability Classification System (MACS), and with spasticity levels ≤2 according to the Modified Ashworth Scale (MAS). Participants were randomly assigned to either an intervention or a control group. Both groups received a standardized physiotherapy and occupational therapy program five days a week for four weeks. In addition to the standard care, the intervention group performed daily 45-minute sessions of core stabilization exercises.

Outcome measures included the Pediatric Berg Balance Scale (PBBS) and the Trunk Control Measurement Scale (TCMS) for evaluating balance, and the Box and Block Test (BBT) and the Assisting Hand Assessment (AHA) for assessing upper extremity function. Assessments were conducted at baseline and post-intervention. The study hypothesized that children receiving core stabilization exercises in addition to standard therapy would show greater improvements in balance and upper extremity function compared to those receiving standard therapy alone.

ELIGIBILITY:
Inclusion Criteria: Who had no other medical conditions that could affect the evaluation and had not had surgery in the past six months.

Exclusion Criteria: Children with severe intellectual disability, muscle contractures or bone deformities, visual impairments, uncontrolled seizures, other neuromuscular diseases, spinocerebellar ataxia, autism spectrum disorder, or communication disorders, as well as children diagnosed with hyperactivity and attention deficit disorder, were excluded from the evaluation. Patients classified as level IV or V according to the Gross Motor Function Classification System (GMFCS), with a spasticity level of 3 or higher according to the Modified Ashworth Scale (MAS), and classified as level IV or V according to the Manual Ability Classification System (MACS) were not included in the study. -

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | From enrollment to the end of treatment at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University,Vocational School of Kocaeli Health Services, Kocaeli University, Umuttepe Campus, 41380, Kocaeli, TURKEY., Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kucuk KE, Cekmece C. The Effect of Core Stabilization Exercises on Upper Extremity Function and Balance in Children with Cerebral Palsy: A Randomized Controlled Trial. Healthcare (Basel). 2025 Jun 17;13(12):1454. doi: 10.3390/healthcare13121454. PMID 40565481